CLINICAL TRIAL: NCT03046446
Title: An Open-label Study to Assess the Safety of Repeat Administration of FX006 to Patients With Osteoarthritis of the Knee
Brief Title: Study to Assess the Safety of Repeat Administration of FX006 Administered to Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FX006-2016-011
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee; Pain; Steroid; Intra-articular; Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — FX006

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FX006 32 mg (Experimental): Single intra-articular injection
  Interventions: Drug: FX006 32 mg

INTERVENTIONS:
Drug: FX006 32 mg — Single intra-articular injection

SUMMARY:
This is an Open-label Study to Assess the Safety of Repeat Dose of FX006 Administered to Patients with Osteoarthritis (OA) of the Knee

DETAILED DESCRIPTION:
This study is an open-label, repeat administration design of 32 mg FX006. The study will be conducted in male and female patients ≥ 40 years of age with symptomatic OA of the knee.

Eligible patients will be offered participation to receive an initial intra-articular (IA) injection of FX006 administered to the index knee at Day 1.

Patients who receive an initial injection of FX006 will return at Weeks 4 and 8 before being evaluated at 12, 16, 20 and 24 weeks for repeat administration. At the first evaluation where the patient has been determined to meet repeat administration eligibility criteria, the patient will be eligible to receive a second IA injection of FX006.

Patients who are eligible to receive a second injection will be evaluated for a total of 52 weeks post initial injection at: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52, regardless of the time at which they receive their second injection. In addition, X-rays will be completed at Screening and Week 52 or End of Study (EOS) for assessment of safety.

Patients that do not benefit from the initial treatment as determined by evaluation at Week 12 will complete the study at the Week 12 follow-up visit.

Patients who are not eligible for a second injection of FX006 after evaluation at Weeks 12, 16, 20, and 24 will complete the study at the Week 24 follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female ≥ 40 years of age
* Symptoms associated with OA of the index knee for ≥ 6 months prior to Screening
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA
* Kellgren-Lawrence (KL) Grade 2, 3 or 4 in the index knee based on X-ray performed during Screening
* Qualifying score for WOMAC A at Screening and Day 1/Baseline
* Index knee pain for >15 days over the last month (as reported by the patient)
* Body mass index (BMI) ≤ 40 kg/m2
* Ambulatory and in good general health
* Willingness to abstain from use of protocol-restricted medications during the study

Exclusion Criteria:

* Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* History of infection in the index knee joint
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee within 1 month of Screening
* Presence of surgical hardware or other foreign body in the index knee
* Unstable index knee joint (such as a torn anterior cruciate ligament) within 12 months of Screening
* IA corticosteroid (investigational or marketed) in index knee within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* IV or intramuscular (IM) corticosteroids (investigational or marketed) within 3 months of Screening
* Oral corticosteroids (investigational or marketed) within 1 month of Screening
* Any other IA drug/biologic use within 6 months of Screening or 5 half-lives (whichever is longer) (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy and amniotic fluid injection)
* Prior administration of FX006
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Study Director — Flexion Therapeutics
Locations (17):
- United States (17):
  - Tucson Orthopedic, Tucson, Arizona
  - Dream Team Clinical Research, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - The Andrews Institute, Gulf Breeze, Florida
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - New England Baptist Hospital, Dedham, Massachusetts
  - Rochester Clinical Research, Rochester, New York
  - Duke University, Durham, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - PMG Research of Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spitzer AI, Richmond JC, Kraus VB, Gomoll A, Jones DG, Huffman KM, Peterfy C, Cinar A, Lufkin J, Kelley SD. Safety and Efficacy of Repeat Administration of Triamcinolone Acetonide Extended-release in Osteoarthritis of the Knee: A Phase 3b, Open-label Study. Rheumatol Ther. 2019 Mar;6(1):109-124. doi: 10.1007/s40744-019-0140-z. Epub 2019 Feb 11. PMID 30741382

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FX006 32 mg
Started | 208
Second Injection (1 patient received 2nd injection after week 24 and is not included in the efficacy data analysis.) | 179
Completed at Week 12 | 10
Completed at Week 24 | 6
Completed at Week 52 | 133
Completed | 149
Not Completed | 59
Not completed — Lack of Efficacy | 7
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 14
Not completed — Withdrawn by Investigator/Sponsor | 3
Not completed — Disease Progression (see caveats) | 25
Not completed — Non OA related knee surgery | 1

BASELINE CHARACTERISTICS:
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 170
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 208

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Treatment Emergent Adverse Events (TEAEs) in Patients With Symptomatic Osteoarthritis (OA) of the Knee Who Received Two Doses of 32 mg FX006
Description: Analyses of adverse events (AE) were performed for events considered treatment-emergent (TE) in patients who received two doses of 32 mg FX006. TE was defined as any AE with onset after administration of the 1st dose of study drug or any event present at baseline but worsened in intensity through the study. Severity was graded by the PI using the Common Terminology Criteria for AEs Version 4.0. Grading went from Grade 1 (Mild) to Grade 5 (Death Related to AE).
Time Frame: Up to 52 Weeks
Population: Received 2 doses of FX006
Measure: Number; unit: TEAEs
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 179
TEAEs | 336

2. Other Pre Specified Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A Pain Subscale
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. WOMAC A is the independent sub-scale for pain that is comprised of 5 questions.
  WOMAC A was administered at each visit from screening through Week 52/EOS.
Time Frame: 12 Weeks Post Each FX006 Administration
Population: Participants who received a repeat administration of FX006 at weeks 12, 16, 20 or 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 178
score on a scale
  Baseline - First Administration | 2.15 (0.580)
  4 Weeks Post First Administration | 0.66 (0.581)
  8 Weeks Post First Administration | 0.83 (0.663)
  12 Weeks Post First Administration | 1.29 (0.765)
  Baseline - Second Administration | 2.00 (0.639)
  4 Weeks Post Second Administration | 0.83 (0.667)
  8 Weeks Post Second Administration | 0.93 (0.691)
  12 Weeks Post Second Administration | 1.28 (0.862)

3. Other Pre Specified Outcome: WOMAC B Stiffness Subscale
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. WOMAC B is the independent sub-scale for stiffness that is comprised of 2 questions.
  WOMAC B was administered at each visit from screening through Week 52/EOS.
Time Frame: 12 Weeks Post Each FX006 Administration
Population: Participants who received a repeat administration of FX006 at weeks 12, 16, 20 or 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 178
score on a scale
  Baseline - First Administration | 2.48 (0.715)
  4 Weeks Post First Administration | 0.74 (0.662)
  8 Weeks Post First Administration | 0.90 (0.749)
  12 Weeks Post First Administration | 1.41 (0.936)
  Baseline - Second Administration | 2.16 (0.824)
  4 Weeks Post Second Administration | 0.88 (0.764)
  8 Weeks Post Second Administration | 0.99 (0.837)
  12 Weeks Post Second Administration | 1.40 (1.007)

4. Other Pre Specified Outcome: WOMAC C Function Subscale
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. WOMAC C is the independent sub-scale for function that is comprised of 17 questions.
  WOMAC C was administered at each visit from screening through Week 52/EOS.
Time Frame: 12 Weeks Post Each FX006 Administration
Population: Participants who received a repeat administration of FX006 at weeks 12, 16, 20 or 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 178
score on a scale
  Baseline - First Administration | 2.18 (0.613)
  4 Weeks Post First Administration | 0.66 (0.593)
  8 Weeks Post First Administration | 0.87 (0.711)
  12 Weeks Post First Administration | 1.28 (0.801)
  Baseline - Second Administration | 1.96 (0.692)
  4 Weeks Post Second Administration | 0.85 (0.685)
  8 Weeks Post Second Administration | 0.96 (0.699)
  12 Weeks Post Second Administration | 1.31 (0.845)

5. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) QOL Subscale
Description: KOOS is a participant (patient)-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury and also consequences of primary osteoarthritis (OA). It holds 42 items in five separately scored sub-scales: KOOS Pain, KOOS Symptoms, Function in daily living, Function in Sport and Recreation, and knee-related Quality of Life (KOOS QOL). Only KOOS QOL sub-scale (Q1-Q4) was used in this study.
  A Likert scale is used and all items have five possible answer options scored from 0 (No Problem) to 4 (Extreme Problems). Each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems. Higher scores indicate a better quality of life.
  KOOS was administered at study visits from BL/Day 1 through week 52.
Time Frame: Up to 12 Weeks Post Each FX006 Administration
Population: Participants who received a repeat administration of FX006
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006 32 mg
Number analyzed (Participants) | 178
score on a scale
  Baseline - First Administration | 28.92 (15.872)
  4 Weeks Post First Administration | 58.06 (22.049)
  8 Weeks Post First Administration | 55.34 (21.791)
  12 Weeks Post First Administration | 46.08 (20.860)
  Baseline - Second Administration | 33.47 (17.270)
  4 Weeks Post Second Administration | 54.85 (20.927)
  8 Weeks Post Second Administration | 50.92 (20.781)
  12 Weeks Post Second Administration | 46.52 (23.274)

ADVERSE EVENTS:
Time Frame: For patients who received a single injection, adverse events were collected following intra-articular (IA) administration through the final study visit at week 24. For patients who received a repeat injection, adverse events were collected following first IA administration through the final study visit at week 52.
Arm/Group | FX006 32 mg
All-Cause Mortality (participants affected / at risk) | 0/208
Serious Adverse Events (participants affected / at risk) | 4/208
Other Adverse Events (participants affected / at risk) | 93/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FX006 32 mg (N=208)
Pancreatitis (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FX006 32 mg (N=208)
Influenza (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 16
Ligament sprain (Injury, poisoning and procedural complications) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 60
Back pain (Musculoskeletal and connective tissue disorders) | 8
Joint crepitation (Musculoskeletal and connective tissue disorders) | 7
Joint effusion (Musculoskeletal and connective tissue disorders) | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9

LIMITATIONS AND CAVEATS:
Disease progression defined as response to first and second injections but loss of effect sometime after the response to the second injection. All discontinuations because of disease progression occurred ≥ 12 weeks after the second injection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT03046446/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT03046446/SAP_001.pdf